CLINICAL TRIAL: NCT03558945
Title: Clinical Trial to Evaluate Safety and Effect of Personalized Neoantigen Vaccine for Pancreatic Tumor Following Surgical Resection and Adjuvant Chemotherapy
Brief Title: Clinical Trial on Personalized Neoantigen Vaccine for Pancreatic Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anda Biopharmaceutical Development (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP03
Record Dates: First submitted 2018-05-24; First posted 2018-06-15 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Tumor
Keywords: pancreatic tumor; neoantigen; vaccine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized neoantigen vaccine (Experimental): Patients will receive radical resection surgery and at least one circle of post-operative chemotherapy. After chemotherapy, personalized neoantigen vaccines will be administered subcutaneously.
  Interventions: Biological: Personalized neoantigen vaccine

INTERVENTIONS:
Biological: Personalized neoantigen vaccine — Patients will have complete resection of primary tumor without preoperative chemotherapy. Patients will receive postoperative chemotherapy and subsequently personalized vaccines on days 1, 4, 8, 15, 22 (priming phase) and weeks 12, 20 (boosting phase). Personalized vaccines will consist of several distinct peptides (the dose is 0.3 mg/peptide) that are grouped into 2-4 pools and 0.5 mg of poly-ICLC as the adjuvant for each pool. Injection sites will be 2-4 separate sites of the subject's thighs.

SUMMARY:
This clinical trial is to evaluate the safety and impact on prognosis of personalized neoantigen peptide-based vaccines, which are based on next-generation sequencing and major histocompatibility complex affinity prediction algorithm, in patients with pancreatic ductal adenocarcinoma. The hypothesis of this study is that personalized neoantigen vaccines will be safe and can systemically elicit measurable neoantigen-specific immunologic responses in patients. Participants will receive complete macroscopic resection of primary tumor, standard adjuvant chemotherapy and subsequently personalized neoantigen vaccines.

DETAILED DESCRIPTION:
This is a single-center, open-label Phase Ib clinical trial. In this trial, adult subjects with pancreatic ductal adenocarcinoma who have completed resection of the primary tumor and who have not undergone preoperative chemotherapy will be enrolled in the study. Eligible enrolled patients all will undergo tumor resection and all receive adjuvant chemotherapy prior to preparation of the personalized neoantigen vaccine. After the chemotherapy finish, subsequently patients will receive a priming immunization with five doses of the personalized neoantigen vaccine over one month and a boosting immunization with two doses three months later. This clinical trial will examine the safety and effect of the personalized neoantigen vaccine when given at several different time points and will examine the participant's peripheral blood cells for signs that the vaccine induces immunologic responses. Finally we will establish the typical flow to assess efficiency and safety of vaccines according to the different reactivity of patients, as a result, to explore the most suitable practical approaches for applying personalized pancreatic tumor vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis of pancreatic ductal adenocarcinoma
2. Aged ≥20 and ≤75
3. Male or not pregnant women
4. Undergone radical resection (R0 status of resection margins [no cancer cells within 1 mm of all resection margins])
5. No serious underlying disease, Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. No chemotherapy or radiotherapy before resection surgery
7. No significant cardiac, lung, liver, kidney, and bone marrow insufficiency
8. No HIV or syphilis infection
9. Signing informed consent

Exclusion Criteria:

1. Poor postoperative situation
2. Obvious organ dysfunction
3. Radiographically confirmed recurrence or metastasis within 180 days after the surgery
4. Unstable angina pectoris, symptomatic congestive heart failure, severe arrhythmias, Myocardial infarction in the past 6 months, and prolonged QT interval (> 450ms)
5. Previous malignant tumors other than pancreatic cancer
6. Cannot be follow up
7. Participating in other clinical trials
8. Without chemotherapy after resection surgery

Exit criteria:

1. Missed within one month after surgery or not follow-up as required
2. Patient's own willingness to withdraw
3. Concurrent disease or severe adverse events
4. Protocol violations
5. Administrative reasons

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and grades of adverse events as assessed by CTCAE v5.0 | From the first dose of vaccination through 2 years after the surgery
  Safety will be assessed by the rate of grade 3 or worse adverse events (graded according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0).

SECONDARY OUTCOMES:
Recurrence-free survival | From the date of resection surgery until the date of the first confirmed tumor recurrence or date of death from any cause or date of study completion, whichever came first, assessed up to 6 years.
  The time between resection surgery and the tumor recurrence (radiological assessment of disease status according to RECIST1.1 criteria).
Overall survival | From the date of resection surgery until the date of death from any cause or date of study completion, whichever came first, assessed up to 6 years.
  The time between resection surgery and the death (any cause).
Serum CA19-9 or CA72-4 levels | From the date of resection surgery until the date of last documented examination of CA19-9 and CA72-4 or date of study completion, whichever came first, assessed up to 6 years.
  The rate of patients without the abnormal elevation of the serum CA19-9 (Cancer Antigen 19-9) or CA72-4 (Cancer Antigen 72-4) levels will be assessed during the vaccination and post-treatment follow-up.

OTHER OUTCOMES:
Levels of interferon-γ responses in peripheral blood mononuclear cells | From the date of first dose of vaccination through 264 days after the first dose of vaccination.
  Ex vivo Enzyme-linked Immunospot assay will be performed to detect the levels of interferon-γ responses of the neoantigen peptides in the stimulation of peripheral blood mononuclear cells. Data will be presented as the ratio of the adjusted spot-forming count of peptide stimulation to the corresponding non-stimulated negative control.
Percentages of immune cell populations in peripheral blood during the vaccination | From the date of first dose of vaccination through 264 days after the first dose of vaccination.
  The percentages of immune cells including natural killer (NK) cells, T cells, B cells, macrophages, monocytes, dendritic cells and granulocytes as well as their subtypes will be detected in the peripheral blood of patients during the vaccination. The percentages of specific T-cell or B-cell clonotypes will also be detected during the vaccination. Ten-color flow cytometry and single-cell transcriptome sequencing will be performed to evaluate the percentage of the immune cell populations. Single-cell T/B-cell repertoire sequencings will be performed to profile the expansion of T-cell or B-cell clonotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Doctor, Principal Investigator — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China